CLINICAL TRIAL: NCT01786759
Title: Hepatic Function and Bile Acid in Preterm Infants Receiving Parenteral Lipids Emulsion
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Wei Cai, vice-president, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HFBA
Record Dates: First submitted 2013-02-06; First posted 2013-02-08 (Estimated); Last update posted 2013-02-08 (Estimated); Status verified 2013-02

CONDITIONS: Preterm Infants
Keywords: lipids; preterm infants; parenteral nutrition; liver function
MeSH Terms: conditions — Hyperphagia | interventions — ClinOleic; soybean oil, phospholipid emulsion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- LCT lipid emulsion (Active Comparator): the LCT lipid emulsion is Intralipid
  Interventions: Drug: ClinOleic; Drug: Intralipid
- Olive oil lipid emulsion (Experimental): the olive oil lipid emulsion is ClinOleic
  Interventions: Drug: ClinOleic; Drug: Intralipid

INTERVENTIONS:
Drug: ClinOleic — the lipid of all-in-one, 0.5-3.5g/kg.d
Drug: Intralipid — the lipid of all-in-one, 0.5-3.5g/kg.d

SUMMARY:
The etiology of parenteral nutrition-associated cholestasis(PNAC)although elusive is thought to be multifactorial, and proposed theories also include problems arising from lipid emulsions, leading us to explore alternative products available elsewhere.So we compare the different fat emulsion, and want to see if the olive oil lipid emulsions can improve hepatic tolerance in preterm infant.

DETAILED DESCRIPTION:
Parenteral nutrition (PN) has been widely and successfully used in the pediatric population for more than 40 years, the most serious and significant life-threatening complication today continues to be parenteral nutrition-associated cholestasis(PNAC). Parenteral nutrition-associated cholestasis is indeed the most worrisome complication because it is difficult to treat and may progress to eventual cirrhosis and liver failure namely parenteral nutrition-associated liver disease (PNALD).

Two types of lipid emulsions are currently used for adult as well as pediatric patients: one lipid emulsions prepared from soybean oil that are composed of long-chain triacylglycerols (LCTs), and the other lipid emulsions composed of 50% medium-chain triacylglycerols (MCTs) and 50% LCT soybean oil. A new lipid emulsion prepared from a mixture of soybean oil and olive oil contains only LCTs and has a lower proportion (20%) of polyunsaturated fatty acids(PUFAs)and 60% monounsaturated fatty acids (MUFAs). So we compare the different fat emulsion, and want to see if the olive oil lipid emulsions can improve hepatic tolerance in preterm infant.

ELIGIBILITY:
Inclusion Criteria:

* Infants of both genders
* Hospitalized
* The parent of the infant agreed to participate by signing an informed consent form
* Infants admitted hospital within 72 hours after birth(gestational age<37 weeks)
* Birth weight <= 2000g
* No PN support contraindications
* Parenteral nutrition for 14 days or more
* The parent of the infant is to sign an informed consent form prior to enrollment

Exclusion Criteria:

* Receiving PN before screening
* Enteral nutrition(EN)caloric>10%
* Obstruction jaundice
* Suspected or identified biliary tract atresia
* Neonatal hepatitis
* Infants with liver markers >2 times normal levels
* Infants with renal markers >2 times normal levels
* Congenital metabolic situations
* Identified as having major chromosomal disease
* Cytomegaoviyns(CMV), virus hepatitis and syphilis infection
* Congenital or acquired immune deficiency

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2012-10; Primary Completion 2013-05 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
liver function | Change from Baseline in fatty acid at 7 days and 14 days
  Total Bile Acid(TBA),alanine aminotransferase(ALT),aspartate aminotransferase(AST),alkaline phosphatase(AKP),γ-glutamyl transpeptidase(GGT),total bilirubin(Tbi),Direct bilirubin(Dbi)

SECONDARY OUTCOMES:
bile acid | Change from Baseline in fatty acid at 7 days and 14 days
  cholic acid,deoxycholic acid,Chenodeoxycholic Acid,ursodeoxycholic acid,lithocholic acid,et al.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Cai, PhD, Study Chair — Xin Hua Hospital; Ying Wang, PhD, Principal Investigator — Xin Hua Hospital, School of Medicine, Shanghai Jiao Tong University
Locations (1):
- Xinhua hospital, Shanghai, Shanghai Municipality, China